CLINICAL TRIAL: NCT03264768
Title: Endoscopic Long Volume Reduction by Endobronchial Valves in Belgium
Acronym: BEVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Wim Janssens, Clinical Professor, KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s60207
Record Dates: First submitted 2017-08-01; First posted 2017-08-29 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: valves; Chronic Obstructive Pulmonary Disease; endoscopic long volume reduction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Pneumonectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Other): standard care in case collateral ventilation is observed (by Chartis) with 3 months physical activity tele coaching between 3 and 6 months post allocation.
  Interventions: Behavioral: physical activity tele coaching; Procedure: Lung volume reduction surgery (LVRS)
- Endobronchial valves (Experimental): Endobronchial valves in case collateral ventilation is absent (by Chartis) with 3 months physical activity tele coaching between 3 and 6 months post intervention.
  Interventions: Device: endobronchial valves; Behavioral: physical activity tele coaching; Procedure: Lung volume reduction surgery (LVRS)

INTERVENTIONS:
Device: endobronchial valves — A ambulatory diagnostic bronchoscopy under general anesthesia will evaluate the presence or absence of collateral ventilation . The targeted lobar airway is temporarily occluded by means of a balloon catheter, which blocks inspiratory flow but allows expiratory flow, in order to assess whether the air flow gradually declines to zero, meaning absence of collateral ventilation. Only in case collateral ventilation is excluded, a therapeutic bronchoscopy will be scheduled to insert the one-directional endobronchial valves in the targeted lobar airways. We will only perform a unilateral intervention during which we will treat one or maximal two lobes at one side.
  Arms: Endobronchial valves
Behavioral: physical activity tele coaching — 3 month physical activity tele coaching intervention consisting of a project tailored smartphone application in combination with a step counter providing direct feedback.
Procedure: Lung volume reduction surgery (LVRS) — Patients not eligible for endoscopic lung volume reduction (or non responders of this intervention) can be referred for surgical lung volume reduction. With this procedure, the most emphysematous parts of the lungs will be surgically removed.

SUMMARY:
This a single center non-randomised non-sham controlled intervention study evaluating the effectiveness and safety of endoscopic lung volume reduction by endobronchial valves

DETAILED DESCRIPTION:
The primary objective of the current study is to explore the effect of targeted lobar endobronchial lung volume reduction in symptomatic patients with severe emphysema and absent collateral ventilation, on lung function, exercise capacity and physical activity. As a secondary objective, changes in physical activity as result of a 3 month activity coaching program delivered between 3 to 6 months post intervention will be investigated. Exploratory objectives are to extend insight in the clinical characteristics of responders and non-responders and to address relationships between lung function response, physical functioning and its impact on inflammation, skeletal and cardiac function. Furthermore, comparison of the effects on lung function, exercise capacity, quality of life and physical activity between endoscopic lung volume reduction and surgical lung volume reduction will be made.

The study will also explore if treatment response can be optimised by an intermediate evaluation with CT scan one month after intervention. Endoscopic evaluation and repositioning of the endobronchial valves will be imposed in case no lober atelectasis is visualised.

.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 - 75 years
* Confluent or destructive heterogeneous emphysema on CT
* Smoking cessation for at least 6m (proven by urinary cotinine levels)
* FEV1 < 60 %predicted, RV > 150 %predicted, TLC > 90 %predicted
* RV/TLC ratio ≥ 0.55
* 6MWD < 450 meter
* mMRC ≥ 2
* Visual estimation of 70% complete fissure between target lobe and adjacent lobe on CT of referring physician
* LABA-LAMA bronchodilator therapy as a minimum therapy
* Able to sign informed consent

Exclusion Criteria:

* Homogenous emphysema
* PaCO2 > 60 mmHg with ambient air
* PaO2 < 45 mmHg with ambient air
* Previous LVRS, lung transplantation, lobectomy
* TLCO or FEV1 < 20% predicted
* Significant pulmonary hypertension (PaPsyst > 50 mm Hg)
* Heart failure with reduced EF (< 40%)
* 6MWD < 100 meter
* BODE index ≥ 7 and eligible for transplantation
* Active cancer
* Life expectancy < 3 months
* Significant lung disease other than COPD/emphysema
* Unable to comply with study procedures

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
response rate of FEV1 at 3 months post intervention | 3 months
  proportion of patients with a minimal change of FEV1 > 100 ml

SECONDARY OUTCOMES:
response rate on SGRQ at 3 months and 6 months post intervention | 3 months and 6 months post intervention
  proportion of patients with a minimal change of -4 points on SGRQ
response rate on 6 minutes walking distance (6MWD) at 3 months and 6 months post intervention | 3 months and 6 months post intervention
  proportion of patients with a minimal improvement of 30 meters on 6MWD
response rate on residual volume (RV) at 3 months and 6 months post intervention | 3 months and 6 months post intervention
  proportion of patients with a minimal reduction of 400 ml on residual volume
response rate on FEV1 at 6 months post intervention | 6 months
  proportion of patients with a minimal change of FEV1 > 100 ml
response rate on Transitional dyspnee index (TDI) at 3 months and 6 months post intervention | 3 months and 6 months post intervention
  proportion of patients with a minimal change of -1 point on TDI

OTHER OUTCOMES:
Change in FEV1 (liters), FVC (liters), RV (liters), TLC (liters) at 3 and 6 months post intervention | 3 months and 6 months post intervention
  Absolute difference from baseline values (liters)
Change in RV/TLC ratio (%) at 3 and 6 months post intervention | 3 months and 6 months post intervention
  Absolute difference from baseline values (%)
Change in 6MWD (meters) at 3 and 6 months post intervention | 3 months and 6 months post intervention
  Absolute difference from baseline values (meters)
Change in physical activity at 3 months post intervention | 3 months post intervention
  Absolute difference in stepcounts per day (n) from baseline values
Change in ProActive clinical visit questionnaire | 3 months post intervention
  Absolute difference in points from baseline values
Change in BODE index | 3 months and 6 months post intervention
  Absolute difference in points from baseline values
changes in physical activity between 3 and 6 months of follow up (telecoaching period) | 3 months - 6 months post allocation
  Absolute difference in stepcounts per day (n) 3 months - 6 months post allocation
changes in ProActive clinical visit questionnaire between 3 and 6 months of follow up (telecoaching period) | 3 months - 6 months post allocation
  Absolute difference in points 3 months - 6 months post allocation
Comparing change in FEV1 (liters), FVC (liters), RV (liters), TLC (liters) at 3 and 6 months post EBV and LVRS | 3 months and 6 months post intervention (endoscopic or surgical)
  Absolute difference from baseline values (liters) for both interventions
Comparing change in 6MWD at 3 and 6 months post EBV and LVRS | 3 months and 6 months post intervention (endoscopic or surgical)
  Absolute difference from baseline values (meters) for both interventions
Comparing change in physical activity at 3 and 6 months post EBV and LVRS | 3 months and 6 months post intervention (endoscopic or surgical)
  Absolute difference from baseline values (amount of steps per day) for both interventions
Comparing change in SGRQ at 3 and 6 months post EBV and LVRS | 3 months and 6 months post intervention (endoscopic or surgical)
  Absolute difference from baseline values for both interventions

CONTACTS AND LOCATIONS:
Overall Officials: Wim Janssens, MD, Principal Investigator — University hospital Leuven, Belgium; Dooms Christophe, MD, Principal Investigator — University Hospial Leuven, Belgium
Locations (1):
- UZ Leuven, Leuven, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No